CLINICAL TRIAL: NCT07182448
Title: Interaction of Hypoxia and Kynurenine Pathway in Periodontal Inflammation
Brief Title: Hypoxia and Kynurenine Pathway in Periodontal Inflammation
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Ankara University (Other)
Responsible Party: Principal Investigator, Nur Balci, DDs, PhD, Clinical Prof, Istanbul Medipol University Hospital
Other Study IDs: 1124
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Periodontitis; Diagnose Disease
Keywords: hypoxia; kynurenine; oxidative stress; periodontitis; tryptophan
MeSH Terms: conditions — Periodontitis; Hypoxia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Saliva and serum collection of patients and samples molecules analysis: Saliva and serum collection of patients and samples molecules analysis Saliva and serum sampling Saliva were collected to analyze the selected markers as unstimulated samples during the early hours of the day. The saliva was centrifuged and then transferred into Eppendorf tubes. Venous puncture was performed after saliva collection and 10 mL of blood samples were collected by qualified staff from each participant. Saliva and serum were then stored at -80 °C until analysis.
  Interventions: Other: Saliva and serum sampling
- Salivary and serum TNF-α, HIF-1α, 8-OhdG , KYN, TRP observation: Salivary and serum tumor necrosis factor-alpha (TNF-α), hypoxia-inducible factor-1 alpha (HIF-1α) and 8-hydroxy-2'-deoxyguanosine (8-OhdG) levels were evaluated by ELISA, and salivary and serum KP metabolites were evaluated by liquid chromatography-mass spectrometry.
  Interventions: Other: Saliva and serum sampling

INTERVENTIONS:
Other: Saliva and serum sampling — Saliva were collected to analyze the selected markers as unstimulated samples during the early hours of the day. The saliva was centrifuged and then transferred into Eppendorf tubes.
  Venous puncture was performed after saliva collection and 10 mL of blood samples were collected by qualified staff (MFD) from each participant. Saliva and serum were then stored at -80 °C until analysis.

SUMMARY:
The kynurenine pathway (KP), the primary route for tryptophan (TRP) metabolism, is activated during inflammation and hypoxic conditions, contributing to immune dysregulation and oxidative stress. the interconnected roles of hypoxia, KP activation, and oxidative stress in periodontitis have not been comprehensively investigated.The aim of this study was to determine the role of the kynurenine (KYN) pathway and hypoxia in periodontal inflammation, as well as their association with periodontal clinical parameters.

DETAILED DESCRIPTION:
Systemically healthy 23 stage III, grade B periodontitis patients and 22 periodontally healthy individuals were included in this study. Salivary and serum tumor necrosis factor-alpha (TNF-α), hypoxia-inducible factor-1 alpha (HIF-1α) and 8-hydroxy-2'-deoxyguanosine (8-OhdG) levels were evaluated by ELISA, and salivary and serum KP metabolites were evaluated by liquid chromatography-mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy
* clinical diagnosis of periodontitis
* clinical diagnosis of periodontal health

Exclusion Criteria:

* decline to participate and being under 18 & over 65 years of age;
* having any systemic inflammatory diseases such as diabetes, rheumatoid arthritis, or systemic conditions, including immunodeficiency syndrome, cardiovascular disorders, or hepatic disorders;
* the use of antibiotics and/or anti-inflammatory nonsteroidal anti-inflammatory drugs within 3 months preceding the study;
* having nonsurgical periodontal treatment (previous 6 months);
* having surgical periodontal treatment (previous 12 months);
* having <20 natural teeth excluding the third molars.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Periodontally healthy and stage 3 garde B periodontitis patients were enrolled in this study
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Pocket probing depth | 3 months
  Measurement of the depth of a sulcus or periodontal pocket determined by measuring distance from a gingival margin to the base of the sulcus or pocket with a calibrated periodontal probe
Clinical attachment level | 4 months
  Clinical attachment level (or loss, CAL) is a more accurate indicator of the periodontal support around a tooth than probing depth alone. CAL is measured from a fixed point on the tooth that does not change, the CEJ.
  To calculate CAL, two measurements are needed: distance from the gingival margin to the CEJ and probing depth.
  In recession: probing depth (+) gingival margin to the CEJ (add). In tissue overgrowth: probing depth (-) gingival margin to the CEJ (subtract)
Bleeding on probing | 4 months
  Bleeding on probing referring to bleeding that is induced by gentle manipulation of the tissue at the depth of the gingival sulcus, or interface between the gingiva and a tooth

SECONDARY OUTCOMES:
serum and saliva analyses for selected molecules | 3 months
  ELISA method was used for tumor necrosis factor-alpha (TNF-α), hypoxia-inducible factor-1 alpha (HIF-1α) and 8-hydroxy-2'-deoxyguanosine (8-OhdG) levels evaluation. KP metabolites were evaluated by liquid chromatography-mass spectrometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No